CLINICAL TRIAL: NCT05818930
Title: Assessment of Remote EEG Monitoring (REMI-EEG) in Pediatric Emergency and Adult Critical Care Units
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Epitel, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EpitelUtah22
Record Dates: First submitted 2023-03-07; First posted 2023-04-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- REMI vs Conventional EEG (Other): REMI EEG is as Diagnostically useful as conventional EEG at monitoring patients with suspected seizure events.
  Interventions: Diagnostic Test: REMI

INTERVENTIONS:
Diagnostic Test: REMI — Diagnostic monitoring

SUMMARY:
The goal of this observational study is to compare clinical utility between Remote EEG Monitoring (REMI) and conventional EEG in patients (6 and older) that are undergoing EEG recording in a hospital as part of their routine clinical care. The main question[s] it aims to answer are:

* What is the concurrence of diagnosis made by epileptologist using REMI and full-EEG signals.
* What is the proportion of participants experiencing as seizure at the time of sensor placement, compared between REMI sensor placement and full-EEG placement.

Participants will wear REMI and conventional EEG electrodes at the same time.

DETAILED DESCRIPTION:
Epitel has developed Epilog, a wireless wearable EEG sensor capable of transmitting EEG to a recording, display, and review platform called REMI (Remote EEG Monitoring). Epitel's REMI platform consists of the REMI tablet and four Epilog sensors. The REMI tablet requires connection to secure WiFi access, and Emergency Department and Intensive Critical Care's IT to open access to http://remi.epitel.com. The four epilog sensors communicate directly with the REMI tablet via Bluetooth connection. REMI synchronizes four Epilog sensors placed by hospital Emergency Department (ED) or intensive care unit (ICU) staff within minutes of patient arrival, thus allowing patients who are suspected of having encephalopathy to be evaluated quickly and prior to initial treatment. REMI securely transmits EEG data to its cloud server where data are processed in near real time using Persyst® Mobile software. Data can then be remotely reviewed by clinical team members.

The objective of this protocol is to demonstrate clinical utility of the Epilog EEG sensors with the REMI monitoring platform in children age 6 through adults in the pediatric emergency department and neurocritical care unit, respectively. Patients meeting entry criteria will be enrolled by a bedside clinical team member who is trained in Epilog sensor placement and use of the REMI platform. All participants will have four Epilog sensors placed, in addition to the standard of care full-EEG. The bedside clinician will be asked to make a "baseline" diagnosis based only on the clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical EEG has been ordered for suspected seizures
* Age 6 years or older

Exclusion Criteria:

* Cannot undergo EEG recordings because of severe head or other injury that prevents EEG recording.
* Transferred immediately for an operation
* Hemodynamically unstable (SBP less than 90 mmHg) at time of EEG placement
* Inability to place four REMI EEG sensors.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinician's diagnostic impression between REMI and conventional electroencephalograph data. | Through the length of time that a patient is actively monitored using both REMI and a full electroencephalograph (up to 24 hours).
  Concurrence of diagnosis made by epileptologist using REMI and full electroencephalograph signals. (I.e., a comparative count of seizure activity identified by an epileptologist using REMI EEG and using conventional EEG.)

SECONDARY OUTCOMES:
Comparison of time to identify epileptiform EEG signals between REMI and conventional electroencephalograph data. | Time Frame: Through the time of sensor placement for both REMI sensors and a full electroencephalograph (approximately up to one hour).
  Proportion of participants seizing at the time of sensor placement, compared between REMI sensor placement and full electroencephalograph placement. (I.e., a count of seizure activity identified by an epileptologist using REMI EEG before conventional EEG is connected.)

CONTACTS AND LOCATIONS:
Overall Officials: Maija Holsti, MD, MPH, Principal Investigator — University of Utah; Amir M Arain, MD, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Epitel will make this highly-valuable data set available to the wider academic community. This could be done by posting appropriate data on the Epilepsy Ecosystem website: https://www.epilepsyecosystem.org/
  All data collection is performed using the same Epilog Data Dictionary across clinical sites. Each PI and Study Coordinator is trained on the data dictionary reporting. This dictionary follows the Common Data Elements for Epilepsy Mobile Health Systems for which Epitel was a contributing member. The common data elements are meant to standardize to the extent possible all data collection, reporting, and analysis in the epilepsy mobile health space.
Supporting Information: Study Protocol
Time Frame: Requests for data can be submitted starting12 months following study publication and the data may be accessible for up to 24 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement.
URL: http://www.epilepsyecosystem.org/